CLINICAL TRIAL: NCT06528886
Title: V-notes (Transluminal Endoscopic Surgery Through Natural Orifices) Hysterectomy With Regional Anesthesia
Brief Title: V-notes Hysterectomy With Regional Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanliurfa Education and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Seah-2-63
Record Dates: First submitted 2024-07-26; First posted 2024-07-30 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Regional Anesthesia Morbidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- regional anesthesia (Experimental): hysterectomy will be done by V-NOTES under regional anesthesia .
  Interventions: Procedure: hysterectomy by V-NOTES

INTERVENTIONS:
Procedure: hysterectomy by V-NOTES — V-notes is like laparoscopy via the vaginal route.

SUMMARY:
Transluminal endoscopic surgery performed through the natural opening via the vagina is a more comfortable, scarless and less complicated method for patients. This method is similar to laparoscopic surgery and is usually performed under general anesthesia. Regional anesthesia is known to be the most comfortable anesthesia type and has less pain, nausea and vomiting during postoperative recovery. Our aim in this study is to evaluate the results by performing the surgery under regional anesthesia.

ELIGIBILITY:
Inclusion Criteria: Female patient between the ages of 30-70 Preoperative anesthesia evaluation will be evaluated as ASA 1-2 according to the American Society of Anesthesiologists (ASA) physical status Patients who are given a hysterectomy indication due to uterus, cervix and/or adnexal condition and will undergo V-NOTES will be included in the study.

Exclusion Criteria:

Patients contraindicated for spinal anesthesia or pneumoperitoneum, those with a history of tubo-ovarian abscess, deep endometriosis or suspected pelvic adhesions

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — hysterectomy
Enrollment: 17 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
pain score | postoperative first 24 hours
  vas score
complications | postoperative first 24 hours
  bleeding, transfusion

CONTACTS AND LOCATIONS:
Overall Officials: alev esercan, MD, Study Director — Sanliurfa Education and Research Hospital
Locations (1):
- Sanliurfa Education and Research Hospital, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol